CLINICAL TRIAL: NCT06409455
Title: Positive Dementia Caregiving in 30 Days: Randomized Controlled Trial of a Self-guided Automated Online Training Program
Brief Title: Positive Dementia Caregiving: Clinical Trial of an Online Training Program
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Education University of Hong Kong (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Sheung-Tak Cheng, Chair Professor of Psychology and Gerontology, Education University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18622322
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Caregiver Stress Syndrome
Keywords: Family caregiving

STUDY DESIGN:
Intervention Model Description: Randomized parallel group (treatment vs. waitlist control) design
Masking Description: Assessor bias is eliminated by having the assessment instruments administered by the computer in an automated manner, without human involvement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): Caregiver training
  Interventions: Behavioral: Positive Dementia Caregiving in 30 Days
- Waitlist control (Other): Waitlist control
  Interventions: Behavioral: Positive Dementia Caregiving in 30 Days

INTERVENTIONS:
Behavioral: Positive Dementia Caregiving in 30 Days — Based on an evidence-based face-to-face Benefit-Finding Intervention, a computer-delivered web-based program supporting 24/7 access without location restriction, is developed. It is a psychoeducation program with an emphasis on strengthening caregivers' coping capacity through skills training and developing a positive way of looking at caregiving challenges. The program consists of reading materials, illustrated texts, caregivers' testimonies, a chatbot, and several interactive apps to facilitate self-learning at the caregiver's own pace.
  Other Names: Benefit-finding Intervention (Online Version)

SUMMARY:
The goal of this study is to learn if a new online training program is helpful to dementia family caregivers. This online program is fully computerized and supports 24/7 access from any location. The main questions it aims to answer are:

* Does the training program improves the participants' well-being and sense of positive meaning?
* If the program is found to be helpful, does it work through enhancing caregivers' self-belief or getting them to practice positive interpretation of caregiving challenges?

To answer these questions, researchers will compare the online program to a waitlist control.

Participants will:

* Use the intervention (requiring internet access) in a self-guided manner
* Respond to brief questionnaires at the beginning, and 1, 2 and 3 months afterwards

DETAILED DESCRIPTION:
The Benefit-Finding Intervention is a type of caregiver intervention called psychoeducation with psychotherapeutic components. It combines standard topics of psychoeducation (e.g., training of care skills and stress management) with training on thinking style. As implied by the title 'benefit-finding', the training style in focus is the inclination to think alternatively and positively about challenging caregiving situations. In two clinical trials, the Benefit-Finding Intervention was compared with didactic psychoeducational programs but without thought training. This comparison allowed researchers to see if the addition of the benefit-finding component produced improvements over the above those achieved by standard psychoeducation. Results supported the superiority of the Benefit-Finding Intervention, with significantly greater reductions of depression and burden up to 10 months after the termination of the intervention.

A face-to-face intervention is nonetheless labor intensive. It may also cause inconvenience to caregivers who have to find blocks of time to attend the intervention, while making sure the care-recipient is being attended to. Having to travel to receive help is another challenge, especially for rural populations and older caregivers. The limitation of the face-to-face format was further exposed during the pandemic when such meetings were simply impossible. To address these issues, the original Benefit-Finding Intervention has been adapted for computer-automated delivery on a web platform, which is accessible anytime anywhere. The online intervention is not meant to replace traditional manned intervention, but as an alternative service for those who, for various reasons, cannot benefit from traditional interventions or who prefer the flexible, self-guided and self-paced approach offered by this intervention.

ELIGIBILITY:
Inclusion Criteria:

* Having been a dementia caregiver for 3 or more months
* Providing 10 or more hours of care per week
* Scoring 5 or above on the Patient Health Questionnaire-9
* Passing a simple reading comprehension test

Exclusion Criteria:

* Caregiver having participated in any training/therapeutic program on dementia care in the past year
* Care-recipient residing in an institution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2024-12-19 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | baseline, 1 month, 2 months, 3 months
  Patient Health Questionnaire-9; possible scores 0-27, higher = more depressed

SECONDARY OUTCOMES:
Anxiety symptoms | baseline, 1 month, 2 months, 3 months
  Profile of Mood States - Anxiety Subscale, brief version; possible scores 0-24, higher = more anxious
Caregiver burden | baseline, 1 month, 2 months, 3 months
  Zarit Burden Interview, brief version; possible scores 0-24, higher = more burden
Positive aspects of caregiving | baseline, 1 month, 2 months, 3 months
  Positive Aspects of Caregiving Scale, brief version; possible scores 6-30; higher = more positive aspects of caregiving

OTHER OUTCOMES:
Caregiving self-efficacy | 3 weeks
  Revised Scale for Caregiving Self-efficacy, brief version; possible scores 0-100, higher = more self-efficacy
Positive reappraisal coping | 3 weeks
  Brief-COPE, Positive Reframing Subscale; possible scores 2-8, higher = more use of positive reframing

CONTACTS AND LOCATIONS:
Overall Officials: Sheung-Tak Cheng, PhD, Principal Investigator — The Education University of Hong Kong
Locations (1):
- The Education University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Materials will be deposited onto a credible repository.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After study completion
Access Criteria: Open access

REFERENCES:
- [Background] Cheng ST, Chan WC, Lam LCW. Long-Term Outcomes of the Benefit-Finding Group Intervention for Alzheimer Family Caregivers: A Cluster-Randomized Double-Blind Controlled Trial. Am J Geriatr Psychiatry. 2019 Sep;27(9):984-994. doi: 10.1016/j.jagp.2019.03.013. Epub 2019 Mar 26. PMID 31076215
- [Background] Cheng ST, Mak EPM, Kwok T, Fung H, Lam LCW. Benefit-Finding Intervention Delivered Individually to Alzheimer Family Caregivers: Longer-Term Outcomes of a Randomized Double-Blind Controlled Trial. J Gerontol B Psychol Sci Soc Sci. 2020 Oct 16;75(9):1884-1893. doi: 10.1093/geronb/gbz118. PMID 31556447